CLINICAL TRIAL: NCT02142712
Title: Glutaminergic and Histaminergic Pathway Modulation in Acute Ischemic Stroke as an Effective Neuroprotection Strategy.
Brief Title: Histamine Glutamate Antagonism in Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201400353
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Acute Cerebrovascular Accident; Cerebral Edema
Keywords: Ischemic Stroke; Brain Edema; Diphenhydramine; Dextromethorphan; Famotidine
MeSH Terms: conditions — Stroke; Brain Edema; Ischemic Stroke | interventions — Diphenhydramine; Pantoprazole; Famotidine; Dextromethorphan; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pantoprazole (Active Comparator): Pantoprazole intravenous 40mg q daily as part of standard of care for stress ulcer prophylaxis along with current standard of care.
  Interventions: Drug: Pantoprazole
- Famotidine (Active Comparator): Famotidine 40 mg intravenous BID (maximum dose of 80 mg/day) for 4 days as part of standard of care for stress ulcer prophylaxis along with current standard of care.
  Interventions: Drug: Famotidine
- Dextromethorphan (Experimental): Dextromethorphan 60 mg QID orally (maximum dose of 240 mg/day) for 2 days (total of 4 doses) along with current standard of care.
  If the drug can't be given orally, then feeding tube (G-tube, NG Tube or DHT) will be used for drug administration.
  Interventions: Drug: Famotidine; Drug: Dextromethorphan
- Diphenhydramine (Experimental): Diphenhydramine 12.5 mg BID intravenous or 25 mg BID oral for 4 days along with current standard of care.
  Interventions: Drug: Diphenhydramine; Drug: Famotidine

INTERVENTIONS:
Drug: Diphenhydramine — Diphenhydramine 12.5 mg BID intravenous or 25 mg BID oral for 4 days along with current standard of care.
  Other Names: Benadryl
  Arms: Diphenhydramine
Drug: Pantoprazole — Pantoprazole intravenous 40mg q daily as part of standard of care for stress ulcer prophylaxis along with current standard of care.
  Other Names: Protonix
  Arms: Pantoprazole
Drug: Famotidine — Famotidine 40 mg intravenous BID (maximum dose of 80 mg/day) for 4 days as part of standard of care for stress ulcer prophylaxis along with current standard of care.
  Other Names: Pepcid
  Arms: Dextromethorphan; Diphenhydramine; Famotidine
Drug: Dextromethorphan — Dextromethorphan 60 mg QID orally (maximum dose of 240 mg/day) for 2 days (total of 4 doses) along with current standard of care. If the drug can't be given orally, then feeding tube (G-tube, NG Tube or DHT) will be used for drug administration.
  Other Names: Diamox
  Arms: Dextromethorphan

SUMMARY:
Stroke is the 4th leading cause of death in United States with an estimated 1 death every 4 minutes. On average, someone suffers from stroke in United States every 40th second. Stroke recurs in 1 out of 4 stroke patients. About 87% of the strokes are as a result of ischemic insult. The total economic burden from stroke accounts to 38.6 billion dollars per year. Stroke is also one of the leading causes of long term disability. Current stroke therapies concentrate mainly on acute revascularization, sub-acute rehabilitation and secondary prevention.

Neuroprotection is not the mainstay of treatment modality as there are no effective regimen which has satisfied stroke clinicians and researchers. Many neuroprotection agents have shown excellent pre-clinical results but have failed in clinical translation. Thus we need to find new treatments in order to decrease the mortality and morbidity caused by stroke.

The investigators hypothesize that adopting a narrower therapeutic window, with treatment initiation in the first six hours, may demonstrate a positive or significant short and long term neuroprotective effect from NMDA/Glutaminergic or histaminergic antagonism when compared with standard of care.

DETAILED DESCRIPTION:
If the subject decides to take part in this study, the subject will be placed randomly in the treatment group or the standard of care group. This means:

The subject will be given either the treatment drugs with standard of care for stroke or only standard of care. If the subject is placed in the treatment group the subject will be again randomly administered either diphenhydramine oral or through an injection in the vein for 4 days or dextromethorphan tablet orally for 2 days. In the treatment group the subject will receive another drug named famotidine through an injection in vein as a prophylaxis to prevent any gastrointestinal bleeding or ulceration whereas in the standard of care group the subject will receive pantoprazole through an injection in the vein for the same purpose. If the subject cannot take medication orally then we will put a tube through the nose to the subject's stomach or small intestine or we might also put a gastric tube directly into the subject's stomach surgically through a small cut in the belly. The investigators will collect information for the medical charts to include: imaging data, stroke assessments and medical history. A neurological exam will done, called the National Institutes of Health Stroke Scale (NIHSS). It is used to assess the neurologic damage caused by stroke. A Modified Rankin Scale (m-RS) will also be performed and this is a scale used to measure the degree of disability or dependence in the daily activities after a stroke.

The subject will be asked to come for a follow-up at 3 months after the discharge from the hospital and the following will be done:

1. Modified Rankin Scale (m-RS) scores NIH Stroke Scale scores
2. CT or MRI of the head without contrast

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with age ≥18 years and ≤80 years at the time of screening.
2. All Ischemic stroke patients with clinical and or radiological diagnosis.
3. Subjects who have presented to hospital within 6 hours of symptom onset.
4. The subject or his/ her legal representative is willing to undergo informed consent process prior to enrollment into this study.

Exclusion Criteria:

1. Subject with age < 18 years and >80 years at the time of screening.
2. Time of symptom onset cannot be determined.
3. Subject who is pregnant or lactating.
4. Subject who has asthma exacerbations in past 3 months.
5. Subject who has hypersensitivity to dextromethorphan, diphenhydramine or famotidine, or other H2 antagonists or any component of the formulation.
6. Serotonin syndrome.
7. Concurrent administration with or within 2 weeks of discontinuing an MAO inhibitor
8. Subjects with renal or hepatic failure.
9. The subject or legal representative is unable to provide informed consent.
10. The subject is medically unstable to participate in the trial as determined by the principal investigator.
11. The subject has any end stage medical condition as determined by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vishnumurthy S Hedna, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Shands Hospital.
Groups:
- Dextromethorphan: Dextromethorphan- 60 mg QID orally (maximum dose of 240 mg/day) for 2 days (total of 4 doses) + current standard of care
Period: Overall Study
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine | Dextromethorphan
Started | 1 | 1 | 1 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Score
Description: The modified Rankin Scale (m-RS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people after they have suffered a stroke.It is one of the most widely used clinical outcome measure for stroke clinical trials. The score is given according to following scale.
  0- No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 8 days and 3 months from the baseline
Population: The data was not collected since the participants did not come back for follow-ups.
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: National Institutes of Health Stroke Severity (NIHSS) Scale
Description: NIHSS is a tool used by healthcare providers to objectively quantify the degree of impairment caused by a stroke. It is composed of 11 items. Each item scores a specific ability between a score of 0-4. Usually, for each item, a score of 0 indicates normal function in that specific ability, while a higher score indicates some level of impairment. The individual scores from each item are added together to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Time Frame: Baseline
Population: NIHSS data was only collected for the baseline visit, since the participants did not come back for follow-ups.
Measure: Number; unit: NIHSS scale
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Number analyzed (Participants) | 1 | 1 | 1
NIHSS scale | 3 | 3 | 0

3. Primary Outcome: Glasgow Coma Scale (GCS)
Description: Glasgow Coma Scale (GCS) is assessed by physical neurological examination of the subject by a qualified neurologist. GSC is a common scoring system used to describe the level of consciousness in a person following a traumatic brain injury. The initial score correlates with the severity of brain injury and prognosis. It estimates Coma severity based on Eye (4), Verbal (5), and Motor (6) criteria with the following total score of between 3 (indicating deep unconsciousness) and 15 (indicating no issues).
Time Frame: Baseline
Population: Data was collected only for the baseline visit, since the participants did not come back for follow-ups.
Measure: Number; unit: Glasgow Coma Scale
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Number analyzed (Participants) | 1 | 1 | 1
Glasgow Coma Scale | 15 | 15 | 15

4. Primary Outcome: Barthel Index
Description: It is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. It yields a score of 0-20.
  The ten variables addressed in the Barthel scale are:
  1. presence or absence of fecal incontinence
  2. presence or absence of urinary incontinence
  3. help needed with grooming
  4. help needed with toilet use
  5. help needed with feeding
  6. help needed with transfers (e.g. from chair to bed)
  7. help needed with walking
  8. help needed with dressing
  9. help needed with climbing stairs
  10. help needed with bathing
Time Frame: At 3 months from baseline
Population: The data was not collected since the participants did not come back for follow-ups.
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: CT or MRI of Head Without Contrast
Description: MRI of head or CT head done as part of your follow up care at 3 months. This will give us the information about the effect of dextromethorphan effect on the final brain damage from stroke.
Time Frame: At 3 months from baseline
Population: The data was not collected since the participants did not come back for follow-ups.
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to month 3 from the baseline visit
Arm/Group | Famotidine | Pantoprazole | Diphenhydramine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No